CLINICAL TRIAL: NCT01224665
Title: A Phase III Surgical Trial to Evaluate the Benefit of a Standard Versus an Extended Pelvic Lymphadenectomy Performed at Time of Radical Cystectomy for Muscle Invasive Urothelial Cancer
Brief Title: S1011 Standard or Extended Pelvic Lymphadenectomy in Treating Patients Undergoing Surgery for Invasive Bladder Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S1011; SWOG-S1011 (Other Grant/Funding Number: U10CA180888); NCI-2011-02604 (Registry Identifier: NCI)
Record Dates: First submitted 2010-10-19; First posted 2010-10-20 (Estimated); Results first posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Bladder Cancer
Keywords: stage II bladder cancer; stage III bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Active Comparator): therapeutic conventional surgery therapeutic standard lymphadenectomy
  Interventions: Procedure: therapeutic conventional surgery; Procedure: therapeutic standard lymphadenectomy
- Arm II (Experimental): therapeutic conventional surgery therapeutic extended lymphadenectomy
  Interventions: Procedure: therapeutic conventional surgery; Procedure: therapeutic extended lymphadenectomy

INTERVENTIONS:
Procedure: therapeutic conventional surgery — Patients undergo radical cystectomy
Procedure: therapeutic standard lymphadenectomy — Patients undergo standard pelvic lymphadenectomy.
  Arms: Arm I
Procedure: therapeutic extended lymphadenectomy — Patients undergo extended pelvic lymphadenectomy
  Arms: Arm II

SUMMARY:
RATIONALE: Lymphadenectomy may remove tumor cells that have spread to nearby lymph nodes in patients with invasive bladder cancer. It is not yet known whether extended pelvic lymphadenectomy is more effective than standard pelvic lymphadenectomy during surgery.

PURPOSE: This randomized phase II trial is studying standard pelvic lymphadenectomy to see how well it works compared to extended pelvic lymphadenectomy in treating patients undergoing surgery for invasive bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare disease-free survival (DFS) of patients with muscle-invasive urothelial carcinoma of the bladder undergoing radical cystectomy with extended pelvic lymph node dissection (PLND) or standard pelvic lymphadenectomy.

Secondary

* To compare overall survival (OS) of patients randomized to extended PLND versus those randomized to standard pelvic lymphadenectomy.
* To evaluate operative time; whether or not nerve sparing was performed, intraoperative, peri-operative and 90-day morbidity and mortality; length of hospital stay; histology (pure urothelial versus mixed); lymph node counts and lymph node density; adjuvant chemotherapy received; and local and retroperitoneal soft tissue recurrence in patients randomized to extended PLND versus those randomized to standard pelvic lymphadenectomy.
* To collect peripheral blood and two paraffin-embedded blocks of the primary tumor for translational medicine studies, including circulating tumor cells (CTCs) and markers of epithelial and mesenchymal transition, and correlate these findings with pathologic T stage and node metastasis as well as DFS and OS.

OUTLINE: This is a multicenter study. Patients are stratified according to prior neoadjuvant therapy (yes vs no), clinical stage (T2 vs T3 vs T4a), and Zubrod performance status (0-1 vs 2). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo radical cystectomy and standard pelvic lymphadenectomy.
* Arm II: Patients undergo radical cystectomy and extended pelvic lymphadenectomy.

Blood and tumor specimens may be collected periodically for translational studies.

After completion of study therapy, patients are followed up periodically for 6 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed urothelial carcinoma of the bladder

  * Stage T2, T3, or T4a disease

    * No clinical stage consistent with a low-risk of node metastasis (CIS only, T1)
    * No T4b disease (fixed lesion)
  * Disease that requires primary radical cystectomy and lymph node dissection for definitive treatment

    * No laparoscopic surgery
* Predominant urothelial carcinoma with any of the following elements allowed:

  * Adenocarcinoma
  * Squamous cell carcinoma
  * Micropapillary or minor components of other rare phenotype
  * No pure squamous cell carcinoma or adenocarcinoma
* No visceral or nodal metastatic disease proximal to the common iliac bifurcation by 2-view chest x-ray and abdominal-pelvic imaging by computerized tomography or MRI of the abdomen and pelvis
* No intra-operative pelvic lymph node involvement (confirmed by frozen section) at or above the bifurcation of the common iliac vessels in any of the extended template

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-2
* ALT and AST ≤ upper limit of normal (ULN)*
* Alkaline phosphatase ≤ ULN*
* Not pregnant or nursing
* Fertile patients must use an effective contraception
* No other prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or stage I or II cancer from which the patient is in complete remission for the past 5 years
* Medically suitable to undergo cystectomy, in the physician's opinion NOTE: *Levels may be ≥ ULN provided metastatic disease is excluded using dedicated liver imaging, bone scan, or biopsy.

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior partial cystectomy for invasive bladder cancer
* No prior pelvic surgery that would obviate a complete extended lymphadenectomy (e.g., aorto-femoral/iliac bypass)
* Prior neoadjuvant chemotherapy for this cancer allowed provided it has been completed and patient has recovered
* No prior pelvic irradiation

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 658 (Actual)
Dates: Start 2011-11-25 (Actual); Primary Completion 2024-05 (Actual); Study Completion 2024-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seth P. Lerner, MD, Principal Investigator — Baylor College of Medicine
Locations (35):
- United States (29):
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Stanford Cancer Institute, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Louisiana State University Health Sciences Center Shreveport, Shreveport, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Portland Veterans Administration Medical Center, Portland, Oregon
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Baylor Saint Luke's Medical Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Audie L Murphy Veterans Affairs Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
- Canada (6):
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - QEII Health Sciences Centre/Capital District Health Authority, Halifax, Nova Scotia
  - London Regional Cancer Program, London, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - McGill University Department of Oncology, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec

REFERENCES:
- [Derived] Lerner SP, Tangen C, Svatek RS, Daneshmand S, Pohar KS, Skinner E, Schuckman A, Sagalowsky AI, Smith ND, Kamat AM, Kassouf W, Plets M, Bangs R, Koppie TM, Alva A, La Rosa FG, Pal SK, Kibel AS, Canter DJ, Thompson IM Jr; SWOG S1011 Trial Investigators. Standard or Extended Lymphadenectomy for Muscle-Invasive Bladder Cancer. N Engl J Med. 2024 Oct 3;391(13):1206-1216. doi: 10.1056/NEJMoa2401497. PMID 39589370
- [Derived] Kamat AM, Hahn NM, Efstathiou JA, Lerner SP, Malmstrom PU, Choi W, Guo CC, Lotan Y, Kassouf W. Bladder cancer. Lancet. 2016 Dec 3;388(10061):2796-2810. doi: 10.1016/S0140-6736(16)30512-8. Epub 2016 Jun 23. PMID 27345655
- [Derived] Froehner M, Novotny V, Heberling U, Rutsch L, Litz RJ, Hubler M, Koch R, Baretton GB, Wirth MP. Relationship of the number of removed lymph nodes to bladder cancer and competing mortality after radical cystectomy. Eur Urol. 2014 Dec;66(6):987-90. doi: 10.1016/j.eururo.2014.07.046. Epub 2014 Aug 19. PMID 25150172

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 658 participants were enrolled to Step 1 before surgery. 40 of participants did not undergo randomization primarily due to results of their intraoperative assessment. Thus, 618 participants were randomized to Step 2; 315 on the standard LND arm and 303 on the extended LND arm. 26 randomized participants were deemed ineligible. Which leaves a total of 592 randomized and eligible participants, 300 and 292 on the standard and extended LND, respectively.
Groups:
- Standard LND: Active Comparator: Arm I Procedure/Surgery: therapeutic standard lymphadenectomy
- Extended LND: Experimental: Arm II Procedure/Surgery: therapeutic extended lymphadenectomy
Period: Overall Study
Arm/Group | Standard LND | Extended LND
Started | 300 | 292
Completed | 300 | 292
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard LND | Extended LND | Total
Number analyzed (Participants) | 300 | 292 | 592
Age, Continuous [Median (Full Range); unit: years] | 68 [38 to 90] | 69 [37 to 92] | 69 [37 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 56 | 122
  Male | 234 | 236 | 470
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    White | 271 | 265 | 536
    Black | 12 | 10 | 22
    Asian | 7 | 5 | 12
    Other, Multiracial, Unknown | 10 | 12 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Hispanic ethnicity
  Participants
    Hispanic | 6 | 21 | 27
Body Mass Index (BMI) [Median (Full Range); unit: kg/m^2] — The body mass index (BMI) is the weight in kilograms divided by the square of the height in meters.
  kg/m^2 | 27.3 [15.2 to 45.2] | 27.3 [15.6 to 42.8] | 27.3 [15.2 to 45.2]
Zubrod Performance Status of 0 or 1 [Count of Participants; unit: Participants] — Zubrod's performance status scores are assessed on a 5-point scale, with higher numbers indicating greater disability. A score of 0 indicates asymptomatic, a score of 1 indicates symptomatic but completely ambulatory, and a score of 2 indicates ambulatory but unable to carry out work activities.
  Participants
    0-1 | 295 | 288 | 583
    2 | 5 | 4 | 9
Clinical T Stage [Count of Participants; unit: Participants] — Clinical stage of the primary tumor is assessed using AJCC seventh edition, 2010 and is based on TURBT(s) that determined the need for cystectomy, bimanual exam, and cross-sectional imaging. Higher numbers indicate more extensive invasion by the primary tumor. A clinical stage of T2 indicates the tumor invades muscularis propria, T3 the tumor invades perivesical tissue, and T4a indicates the tumor invades the prostatic stoma, uterus, or vagina.
  Participants
    T2 | 213 | 208 | 421
    T3 or T4a | 87 | 84 | 171
Hydronephrosis [Count of Participants; unit: Participants] — Participants who experienced hydronephrosis are reported. Hydronephrosis, also known as obstructive uropathy, is a condition of excess urine accumulation in kidney(s) that causes swelling of the kidneys.
  Participants | 74 | 78 | 152
Mixed Histologic Subtypes [Count of Participants; unit: Participants] — The number of participants with mixed histology (versus pure urothelial histology) are reported.
  Participants | 36 | 12 | 48
Neoadjuvant Chemotherapy [Count of Participants; unit: Participants]
  Any neoadjuvant chemotherapy | 170 | 166 | 336
  Cisplatin-based | 146 | 147 | 293
  Carboplatin-based | 10 | 12 | 22
  Other neoadjuvant chemotherapy | 14 | 7 | 21
  None | 130 | 126 | 256

OUTCOME MEASURES:

1. Primary Outcome: 5-year Disease-free Survival (DFS)
Description: Comparing 5-year disease-free survival (DFS) in participants undergoing radical cystectomy for muscle-invasive urothelial carcinoma of the bladder (UCB) treated with radical cystectomy and extended pelvic lymph node dissection (PLND) compared to radical cystectomy and standard pelvic lymphadenectomy. Disease-free survival is defined as the time from the date of randomization to date of first documentation of relapse/recurrence or death due to any cause. Participants last known to be alive without report of relapse/recurrence are censored at date of last contact. Criteria for recurrence included measurable disease on cross-sectional imaging or plain radiography targeting lung, liver, and bone. If local pelvic recurrence was identified on digital rectal examination, biopsy was required for confirmation. Second primary tumors of the upper urinary tract or retained urethra were not considered to be recurrence.
Time Frame: Duration of treatment and follow-up until death or 6 years after randomization
Measure: Number; unit: percentage of participants
Arm/Group | Standard LND | Extended LND
Number analyzed (Participants) | 300 | 292
percentage of participants | 60 | 56
Statistical Analysis 1: Comparison: Standard LND vs Extended LND; 3-year DFS estimates of 55% among participants undergoing SLND and 65% undergoing ELND were used to estimate the target HR. Assuming exponential DFS distribution, 5 years of enrollment, 3 years of follow-up, and 564 eligible participants, the trial would have 85% power to detect a 28% lower risk of recurrence or death with ELND than SLND; Test type: Superiority; p = 0.45, Log Rank — Using an intention-to-treat analysis, we specified a stratified log-rank test with a one-sided alpha of 0.025; Adjustments were made for the following stratification factors: neoadjuvant chemotherapy, clinical T stage, and Zubrod performance score; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.86 to 1.40] — Adjustments were made for the following stratification factors: neoadjuvant chemotherapy, clinical T stage, and Zubrod performance score

2. Secondary Outcome: 5-year Overall Survival (OS)
Description: Comparing 5-year overall survival (OS) in participants randomized to extended PLND versus those randomized to standard pelvic lymphadenectomy. Overall survival is defined as the time from date of randomization to date of death from any cause. Participants known to be alive are censored at date of last contact.
Time Frame: Duration of treatment and follow-up until death or 6 years after randomization
Measure: Number; unit: percentage of participants
Arm/Group | Standard LND | Extended LND
Number analyzed (Participants) | 300 | 292
percentage of participants | 63 | 59
Statistical Analysis 1: Comparison: Standard LND vs Extended LND; We assumed that the standard lymphadenectomy arm has 5-year survival of 55%, so we had 83% statistical power to detect a hazard ratio of 0.72 (55% vs. 65% survival at 5 years); Test type: Superiority; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.88 to 1.45] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Median Operative Time
Description: Evaluating duration of surgery in participants randomized to extended lymphadenectomy versus those randomized to standard lymphadenectomy.
Time Frame: Duration of surgery
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Standard LND | Extended LND
Number analyzed (Participants) | 300 | 292
hours | 5.3 [4.5 to 6.6] | 5.9 [5.1 to 7.0]

4. Secondary Outcome: Median Days in Hospital
Description: Evaluating duration of post-operative hospital stay in participants randomized to extended lymphadenectomy versus those randomized to standard lymphadenectomy.
Time Frame: From date of operation to 90 days post-operation
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard LND | Extended LND
Number analyzed (Participants) | 300 | 292
days | 6 [5 to 8] | 7 [5 to 9]

5. Secondary Outcome: Use of Nerve Preservation
Description: Evaluating the frequency of nerve sparing surgery in participants randomized to extended lymphadenectomy versus those randomized to standard lymphadenectomy.
Time Frame: Duration of surgery
Population: The overall number of nerve-sparing surgeries performed per arm is reported as well as the numbers for males and females on each arm. The standard LND arm has 234 male participants and 66 females, while the extended LND arm has 236 males and 56 females.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard LND | Extended LND
Number analyzed (Participants) | 300 | 292
Participants
  Male: number analyzed (Participants) | 234 | 236
  Male: No | 143 | 151
  Male: Unilateral | 12 | 9
  Male: Bilateral | 79 | 76
  Female: number analyzed (Participants) | 66 | 56
  Female: No | 60 | 49
  Female: Unilateral | 0 | 0
  Female: Bilateral | 6 | 7
  Overall: No | 203 | 200
  Overall: Unilateral | 12 | 9
  Overall: Bilateral | 85 | 83

6. Secondary Outcome: Lymph Node Counts
Description: Evaluating the number of positive lymph nodes removed during surgery as well as the total number of lymph nodes removed in participants randomized to extended lymphadenectomy versus those randomized to standard lymphadenectomy.
Time Frame: Duration of surgery
Measure: Median (Full Range); unit: number of lymph nodes
Arm/Group | Standard LND | Extended LND
Number analyzed (Participants) | 300 | 292
number of lymph nodes
  Total lymph nodes removed | 24 [6 to 61] | 39 [15 to 94]
  Positive lymph nodes removed | 1 [1 to 16] | 2 [1 to 35]

7. Secondary Outcome: Receipt of Adjuvant Chemotherapy
Description: Evaluating the receipt of adjuvant chemotherapy in participants randomized to extended lymphadenectomy versus those randomized to standard lymphadenectomy. Participants that reported plans to start adjuvant chemotherapy are included in these counts.
Time Frame: From date of operation to 90 days post-operation
Measure: Number; unit: percentage of participants
Arm/Group | Standard LND | Extended LND
Number analyzed (Participants) | 300 | 292
percentage of participants | 11 | 11

8. Secondary Outcome: Frequency of Post-Operative Local Recurrence
Description: Evaluating the frequency of post-operative local and retroperitoneal soft-tissue recurrence in participants randomized to extended lymphadenectomy versus those randomized to standard lymphadenectomy.
Time Frame: From date of operation to 90 days post-operation
Measure: Number; unit: percentage of participants
Arm/Group | Standard LND | Extended LND
Number analyzed (Participants) | 300 | 292
percentage of participants | 9 | 13

9. Secondary Outcome: Post-Operative Morbidity
Description: Evaluating perioperative morbidity (death within 30 days of surgery) and post-operative morbidity (death within 90 days of surgery) in participants randomized to extended lymphadenectomy versus those randomized to standard lymphadenectomy.
Time Frame: From date of operation to 90 days post-operation
Measure: Count of Participants; unit: Participants
Arm/Group | Standard LND | Extended LND
Number analyzed (Participants) | 300 | 292
Participants
  Death within 30 days | 1 | 8
  Death within 90 days | 7 | 19

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow-up until death or 6 years after randomization
Description: 592 eligible participants who received protocol treatment were evaluable for AEs: 300 on the Standard Pelvic Lymph Node Dissection arm and 292 on the Extended Pelvic Lymph Node Dissection arm. Adverse Events (AEs) and Serious Adverse Events (SAEs) are reported by CTCAE Version 4.0.
Arm/Group | Standard LND | Extended LND
All-Cause Mortality (participants affected / at risk) | 117/300 | 124/292
Serious Adverse Events (participants affected / at risk) | 3/300 | 12/292
Other Adverse Events (participants affected / at risk) | 226/300 | 219/292
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard LND (N=300) | Extended LND (N=292)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0
Gastrointestinal fistula (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Death NOS (General disorders) | 0 | 3
Fatigue (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Sudden death NOS (General disorders) | 0 | 1
Sepsis (Infections and infestations) | 2 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 1
Cardiac troponin I increased (Investigations) | 0 | 1
Creatinine increased (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Stroke (Nervous system disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypotension (Vascular disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard LND (N=300) | Extended LND (N=292)
Anemia (Blood and lymphatic system disorders) | 126 | 126
Sinus tachycardia (Cardiac disorders) | 17 | 16
Abdominal pain (Gastrointestinal disorders) | 26 | 26
Constipation (Gastrointestinal disorders) | 23 | 27
Diarrhea (Gastrointestinal disorders) | 20 | 26
Ileus (Gastrointestinal disorders) | 58 | 47
Nausea (Gastrointestinal disorders) | 34 | 34
Vomiting (Gastrointestinal disorders) | 21 | 29
Edema limbs (General disorders) | 16 | 15
Fatigue (General disorders) | 30 | 32
Fever (General disorders) | 26 | 18
Pain (General disorders) | 26 | 22
Sepsis (Infections and infestations) | 12 | 17
Urinary tract infection (Infections and infestations) | 60 | 57
Wound infection (Infections and infestations) | 16 | 23
Wound complication (Injury, poisoning and procedural complications) | 17 | 14
Creatinine increased (Investigations) | 47 | 48
Lymphocyte count decreased (Investigations) | 17 | 15
Platelet count decreased (Investigations) | 29 | 27
Weight loss (Investigations) | 17 | 18
Acidosis (Metabolism and nutrition disorders) | 19 | 12
Anorexia (Metabolism and nutrition disorders) | 19 | 30
Dehydration (Metabolism and nutrition disorders) | 16 | 9
Hyperglycemia (Metabolism and nutrition disorders) | 39 | 28
Hyperkalemia (Metabolism and nutrition disorders) | 11 | 22
Hypoalbuminemia (Metabolism and nutrition disorders) | 21 | 19
Hypocalcemia (Metabolism and nutrition disorders) | 46 | 53
Hypokalemia (Metabolism and nutrition disorders) | 23 | 23
Hypomagnesemia (Metabolism and nutrition disorders) | 22 | 16
Hyponatremia (Metabolism and nutrition disorders) | 25 | 34
Acute kidney injury (Renal and urinary disorders) | 16 | 33
Urinary incontinence (Renal and urinary disorders) | 27 | 14
Surgical and medical procedures-Other (Surgical and medical procedures) | 18 | 25
Hypertension (Vascular disorders) | 22 | 21
Hypotension (Vascular disorders) | 18 | 24
Thromboembolic event (Vascular disorders) | 17 | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-01-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT01224665/Prot_SAP_ICF_000.pdf